CLINICAL TRIAL: NCT06363318
Title: Comparison of Open and Laparoscopic Appendectomy in Pediatric Population
Acronym: Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0003
Record Dates: First submitted 2024-03-30; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Appendicitis Acute
Keywords: Appendicitis; children; laparoscopic appendectomy; open appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: children were randomly divided in two groups. In group A, laparoscopic appendectomy was done. In group B, open appendectomy was done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A laparoscopic appendicectomy (Experimental): In Group A (50 patients) laparoscopic appendicectomy was done
  Interventions: Procedure: Laparoscopic appendicectomy
- Group B open appendicectomy (Active Comparator): In Group B(50 patients) open appendicectomy was done
  Interventions: Procedure: Laparoscopic appendicectomy

INTERVENTIONS:
Procedure: Laparoscopic appendicectomy — In group A laparoscopic appendicectomy was done while in group B Open appendicectomy was done
  Other Names: open appendicectomy

SUMMARY:
Introduction: In the era of minimally invasive surgery, changing trends are towards laparoscopic surgery, first introduced in 1983. Now the preferred operation for children with appendicitis, laparoscopic appendectomy is associated with a reduced risk of wound infection, less postoperative pain and shorter hospital stay as compared to open appendectomy.

Objectives: To compare the outcome of open and laparoscopic appendectomy in children presenting with appendicitis in terms of operative time, postoperative pain, wound infection and hospital stay.

DETAILED DESCRIPTION:
A total of 100 children presenting with acute appendicitis were included in this study, In group A, patients were undergone laparoscopic appendectomy.

In group B, patients were undergone open appendectomy. During surgery, operative time was noted. After surgery, patients were shifted to surgical wards and were followed-up there till discharge. Patients were followed regularly by the researcher for mean post-operative pain at 24 hours. At discharge, hospital stay was noted. Then patients followed up in outpatient department for 10 days for any evidence of wound infection.

ELIGIBILITY:
Inclusion Criteria:

1. Children of age 7-12 years of either gender diagnosed as acute appendicitis
2. pediatric appendicitis score >4

Exclusion Criteria:

1. Children with comorbidities,
2. Perforated appendix
3. Appendicular mass (on clinical examination). -

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Operative time | during surgery
  from time of incision to skin closure
wound infection | 10 days
  It was labelled if there was redness, swelling or pus present at surgical wound site
Hospital stay | 5 days
  It was measured in terms of days required to stay in hospital after surgery. The start time will be the day of operation and end time was the day of discharge from hospital.
Postoperative pain | 48 hours
  It was measured by using visual analogue scale (VAS), which consists of score minimum zero to maximum ten score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sharif, FCPS, Study Chair — King edward Medical University/Mayo Hospital Lahore
Locations (1):
- Muhammad Sharif, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be shared on demand